CLINICAL TRIAL: NCT05461326
Title: All Soft Tissue Quadriceps Tendon Autograft Versus Patellar Tendon Autograft in Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Trial
Brief Title: Quadriceps Tendon Versus Bone Patellar Tendon Bone Autograft ACL Reconstruction RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amit Momaya, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300009203
Record Dates: First submitted 2022-06-28; First posted 2022-07-18 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Disorder; Anterior Cruciate Ligament Injuries
Keywords: quadriceps tendon; bone tendon bone; autograft
MeSH Terms: conditions — Musculoskeletal Diseases; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quad tendon (Active Comparator): ACL graft harvested from the quadriceps tendon
  Interventions: Procedure: Quad tendon
- BTB tendon (Active Comparator): ACL graft harvested from the patellar tendon
  Interventions: Procedure: BTB

INTERVENTIONS:
Procedure: Quad tendon — quadriceps tendon autograft
  Arms: Quad tendon
Procedure: BTB — patellar tendon autograft
  Arms: BTB tendon

SUMMARY:
The choice of autograft for ACL reconstruction continues to be debated. To date, there has only be one completed randomized controlled trial with quad tendon to BTB and the tendon included a bone plug. There has been no study to date comparing an all soft tissue quad tendon to patellar tendon in a randomized controlled trial for ACL reconstruction.

DETAILED DESCRIPTION:
Patients will be recruited from the PI's population base at Highlands Sports Medicine Clinic. Patients in need of an ACL reconstruction will be asked if they are interested in participating in a study comparing BTB and QT autografts by the PI (Dr. Amit Momaya). The benefits and risks of each graft choice will be thoroughly explained. Both graft options are considered equally appropriate management. Interested patients will be screened for eligibility criteria by a research assistant; those matching eligibility will be consented and enrolled in person at the time of the visit.

Patients will be randomized per trial arm assignment to either (i) assignment "0" or (ii) assignment "1". To ensure randomization, a random number generator is used to assign patient numbers and study groups; these assignments are placed with consent information to remain blinded to research personnel and participants until the consent and enrollment process. We anticipate fifty participants per assignment and oen-hundred participants in total. Assignment 0 represents the BTB group. This procedure harvests the patient's middle third of the patella tendon through a single incision for the new ACL graft. When the graft is in place, the graft is secured using a surgical button at the femoral end and a non-absorbable screw at the tibial end. Assignment 1 represents the QT group. This procedure harvests the patient's quadricep tendon through a single incision then utilizes surgical buttons to fix the graft at the tibial and femoral ends. Following enrollment, patients will immediately be notified of their assignment. Patients will also complete KT-1000 manual maximum side-to-side difference measurements . The patient will then be scheduled for ACL reconstruction surgery according to their assignment.

Following reconstruction, standard of care rehabilitation and mobility instructions will be provided. Participants are expected to complete the usual standard of care 2 week, 6 week, 3 month, 6 month, and 9 month postoperative appointments. At the 2 week and 9 month postoperative visits, a routine x-ray will be performed. Aside from a singular KT-1000 measurement and repeated surveys, the patient should not expect any differences in their postoperative visits compared to if they had not participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients younger 65
* ACL insufficiency
* Scheduled to undergo autograft ACL reconstruction
* Appropriate candidate for autograft harvest

Exclusion Criteria:

* <14 or 65>
* Poor autograft candidate (poor tissue quality)
* Multi ligamentous reconstruction (PCL, MCL, or PLC)
* Pregnant or nursing
* High likelihood of remaining non-compliant with physical therapy regimen
* Desire to return to sport prior to 6 months
* Inability to read and write English

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
KT-1000 Arthrometer | Operative Day, 9 Months Post-Operative Clinic Visit
  Measures maximum side-to-side difference of laxity (translation of the tibia in comparison to a fix femur)

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Knee Evaluation Form | 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months post-operative assessment
  The International Knee Documentation Committee Subjective Knee Evaluation Form measures symptoms, function, and sports activity of people with a variety of knee disorders, including ligamentous and meniscal injuries, osteoarthritis, and patellofemoral dysfunction. Normative values have been published for comparison.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months post-operative assessment
  This survey evaluates short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis
Marx Activity Scale | 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months post-operative assessment
  This survey measures activity-related patient-reported outcome.
Single Assessment Numeric Evaluation (SANE) | 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months post-operative assessment
  A rating of the patient's current illness score.
Visual analog scale (VAS) | Post operative day 1, day 2, day 3, week 1, week 2, week 3, week 4, week 6, 3 months, 6 months, 9 months, 12 months, 24 months
  pain rated on a 0-10 scale, 10 being worse
Re-rupture rate | 2 years
  Incidence of rerupture based on clinical and radiographic (MRI) evidence
Short Term Survey (SF-12) | 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months post-operative assessment
  This survey reports the impact of health on a patient's everyday life.
ACL Return to Sport Index (ACL-RSI) | 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months post-operative assessment
  A survey that evaluates patient's psychological readiness as it relates to return to sport.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Momaya, MD, Principal Investigator — Department of Orthopaedic Surgery, University of Alabama at Birmingham
Locations (1):
- UAB Hospital Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No